CLINICAL TRIAL: NCT01277926
Title: Patterns of Care in Hormone-Receptor Positive, Advanced Breast Cancer in Brazil: A Prospective, Observational Study
Brief Title: Patterns of Care in Hormone-receptor Positive, Advanced Breast Cancer
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OBR-DUM-2010/1; D6998L00002 (Other: AstraZeneca)
Record Dates: First submitted 2011-01-12; First posted 2011-01-17 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hormone Receptor Positive, Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize the current patterns of care for patients with hormone-receptor-positive, advanced breast cancer who have failed one prior endocrine therapy in Brazil. To investigate patient-related, disease-related and physician-related characteristics that correlate with the use of either endocrine treatment or chemotherapy in such patients. And to evaluate patients' understanding of the treatment options and their participation in the choice.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast cancer
* Postmenopausal status at the time of enrolment, according to the following definitions:

  * History of bilateral oophorectomy at any age
  * Proven hormonal menopause
* Positive estrogen receptor (ER) and/or progesterone receptor (PR) by immuno
* Failure of one previous endocrine therapy in the adjuvant or metastatic setting
* Use of no more than one previous chemotherapy regimen in the neoadjuvant or adjuvant setting
* Indication to receive chemotherapy or endocrine therapy

Exclusion Criteria:

* Inability to comply with the study protocol
* Use of more than one previous endocrine therapy, regardless of the setting; -- Previous use of chemotherapy for metastatic disease
* Use of neoadjuvant endocrine therapy as the only previous type of endocrine therapy
* Serious medical, surgical or psychiatric comorbidity that, upon investigator's discretion, should preclude participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To assess the treatment choice by the medical oncologist for each patient. | 12 months

SECONDARY OUTCOMES:
To assess determinants of treatment choice | 12 months
To assess the duration of treatment with chemotherapy or endocrine therapy | 12 months
To evaluate the rate of treatment continuation at 6 months | 12 months
  Assess the profile of adverse events with each treatment modality and assess patient participation and understanding in treatment choice

CONTACTS AND LOCATIONS:
Overall Officials: Paulo André Palhares Miranda, Doctor, Study Director — MC Brazil
Locations (6):
- Brazil (6):
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
  - Research Site, Belo Horizonte
  - Research Site, Mogi das Cruzes
  - Research Site, Ribeirão Preto